CLINICAL TRIAL: NCT00522418
Title: An Open Prospective Randomised Long-Term Effectiveness Study, Comparing Best Medical Practice With or Without Adjunctive VNS Therapy in Patients 16 Years and Older With Pharmaco-resistant Partial Epilepsy
Brief Title: Study Comparing Best Medical Practice With or Without VNS Therapy in Pharmacoresistant Partial Epilepsy Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-100
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2012-10

CONDITIONS: Epilepsy; Partial Epilepsy
Keywords: Epilepsy; VNS Therapy
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VNS Therapy (Experimental): VNS Therapy + Best Medical Practice
  Interventions: Device: Vagal Nerve Simulation (VNS) Therapy
- Best Medical Practice (Active Comparator): Best Medical Practice
  Interventions: Drug: Best Medical Practive

INTERVENTIONS:
Device: Vagal Nerve Simulation (VNS) Therapy — VNS Therapy + Best Medical Practice including anti-epileptic drugs
  Arms: VNS Therapy
Drug: Best Medical Practive — Best Medical Practice including anti-Epileptic Drugs
  Arms: Best Medical Practice

SUMMARY:
This is a post-market medical device study. This study will compare best medical practice with or without adjunctive VNS Therapy in patients who are 16 years and older with pharmacoresistant partial epilepsy.

DETAILED DESCRIPTION:
This is a post-market medical device study. This study will compare best medical practice with or without adjunctive VNS Therapy in patients who are 16 years and older with pharmaco-resistant partial epilepsy. The Sponsor, Cyberonics, provides funding for this study. Patients are followed for 26 months, 24 of those months are following the initiation of treatment. No study sites will be permitted to enroll study subjects until Institutional Review Board (IRB)/Ethics Committee (EC) approval has been received.

ELIGIBILITY:
Inclusion Criteria:

* Patient has confirmed partial onset seizures.
* Seizure activity is not adequately controlled by patient's current AED regimen.
* Patient is between 16 and 75 years of age.
* Patient is able to give accurate seizure counts and health outcomes information. Patient is able to complete study instruments with minimal assistance.
* Patient has previously failed at least 3 AEDs in single or combination use.
* During baseline evaluation period, patient should take at least 1 AED.
* Patient should have confirmed epilepsy for a minimum of 2 years.
* Patient's AED regimen is stable for at least 1 month prior to enrolment.
* Patient has at least 1 objective partial onset seizure per month during the 2 months prior to enrolment.
* Patient or legal guardian understands study procedures and has voluntarily signed an informed consent in accordance with institutional and local regulatory policies.

Exclusion Criteria:

* Patient has pseudoseizures or a history of pseudoseizures.
* Patient has idiopathic generalised epilepsy or unclassified epilepsy.
* Patient has ever received direct brain stimulation (cerebella or thalamic) for treatment of epilepsy.
* Patient has had a unilateral or bilateral cervical vagotomy.
* Patient has a history of non-compliance with the completion of a seizure diary.
* Patient has taken an investigational drug within a period of 3 months prior to inclusion.
* Patient is currently using another investigational medical device.
* Patient has a significant cardiac or pulmonary condition currently under treatment.
* Patient has previously undergone brain surgery.
* Patient has a demand cardiac pacemaker, implantable defibrillator, or other implantable stimulator.
* Patient currently lives more than 2 hours from the study site or plans to relocate to a location more than 2 hours from the study site within one year of enrolment in the Study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillippe Ryvlin, MD, Principal Investigator — Hopital Neurologique, Lyon, France; Sophie Leyman, MD, Study Director — Cyberonics Europe
Locations (48):
- Belgium (2):
  - ULB-Hôpital Erasme, Centre de référence pour le traitement de l'épilepsie réfractaire - Neurologie, Brussels
  - UZ Gent, Department of Neurology, 1K12/A, Ghent
- Canada (4):
  - Foothills Hospital, Neurology Department, Calgary, Alberta
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hopital Notre Dame, Montreal, Quebec
  - Montreal Neurological Institute, Clinical Research, Montreal, Quebec
- France (7):
  - CHU Grenoble, Neurology Department, Grenoble
  - Hopital Roger Salengro, Service de Neurologie, Lille
  - Hôpital Neurologique, Untité d'épileptologie, Lyon
  - Hôpital Gui De Chauliac, Service Explorations Neurologiques et Epileptologie, Montpellier
  - Hôpital Sainte-Anne, Service de Neurochirurgie, Paris
  - Service d'exploration des épilepsies, Strasbourg
  - CHU Tours, Service de neurologie, Tours
- Germany (6):
  - Universitätskliniken Bonn, Klinik für Epileptologie, Bonn
  - Universitätsklinik Erlangen, Zentrum für Epilepsie ZEE, Erlangen
  - Klinik der Ernst-Moritz-Arndt-Universität, Neurologische Klinik, Greifswald
  - Epilepsiezentrum Kork, Kehl-Kork
  - Klinikum der Philips-Universität Marburg, Fachbereich, 20 - Medizin / Klinik Neurologie / Epilepsie Zentrum, Marburg
  - Sächsisches Epilepsiezentrum Radeberg, Epilepsiezentrum Kleinwachau, Radeberg
- Italy (10):
  - Azienda Ospedaliero Universitaria - Ospedali Riuniti Umberto I - Lancisi - Salesi, NeuroPsichiatria Infantile, Ancona
  - Universita di Bologna, Clinica Neurologica, Bologna
  - Azienda Ospendaliero-Universitaria, Caressi Dep Neuroscience, Florence
  - Ospedale San Paolo, Centro Epilessia, Milan
  - Universita degli Studi di Cagliari - Policlinico Monserrato, Clinica Neurologica, Monserrato
  - Universita di Pisa, Clinica Neurologica, Pisa
  - Ospedale F. Lotti, NeuroFisioPatalogia, Pontedera
  - Azienda Ospedaliera "Bianchi Melacrino Morelli", Centro Regionale Epilessie, Reggio Calabria
  - Università Cattolica Del Sacro Cuore, Istituto di NeuroChirurgia, Roma
  - Centro Epilessia, Dipartimento di Neuroscienze, Torino
- Netherlands (5):
  - Tergooiziekenhuizen, Dienst Neurologie, Blaricum
  - Medisch Spectrum Twente, Dienst Neurologie, Enschede
  - Stichting Epilepsie Instituut Nederland, Dienst Neurologie, Heemstede
  - Kempenhaeghe, Dienst Neurologie, Oosterhout
  - Medisch Centrum Rijnmond-Zuid, locatie Clara, Dienst Neurologie, Rotterdam
- Spesialsykehuset for Epilepsi, Dep of Neurodiagnostics, Sandvika, Norway
- Spain (5):
  - Hospital Ruber Internacional, Servicio de neurología, Madrid
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Clínico Universitario, Servicio de neurología, Valencia
  - Hospital General de Valencia, Neurology/Neurophisiology, Valencia
  - Hospital General Basico De La Defensa de Valencia, Servicio de neurología, Valencia
- Sweden (4):
  - Institute of Neuroscience and Physiology, Clinical Neuroscience and Rehabilitation, Gothenburg
  - Universitetssjukhuset i Lund, Neurologiska kliniken, Lund
  - Norrlands Universitetssjukhus, Neurocentrum, Umeå
  - Akademiska sjukhuset, Neurocentrum, Uppsala
- United Kingdom (4):
  - Addenbrookes Hospital, Dept of Neurosurgery, Cambridge
  - Walton Centre, Dept of Neurosciences, Clinical Sciences Centre, Fazakerley
  - Kings College Hospital, Dept of Neurosurgery, London
  - National Hospital for Neurology and Neurosurgery, London

REFERENCES:
- [Background] Gilliam F. Optimizing health outcomes in active epilepsy. Neurology. 2002 Apr 23;58(8 Suppl 5):S9-20. doi: 10.1212/wnl.58.8_suppl_5.s9. PMID 11971128
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Sillanpaa M, Jalava M, Kaleva O, Shinnar S. Long-term prognosis of seizures with onset in childhood. N Engl J Med. 1998 Jun 11;338(24):1715-22. doi: 10.1056/NEJM199806113382402. PMID 9624191
- [Background] Mattson RH, Cramer JA, Collins JF, Smith DB, Delgado-Escueta AV, Browne TR, Williamson PD, Treiman DM, McNamara JO, McCutchen CB, et al. Comparison of carbamazepine, phenobarbital, phenytoin, and primidone in partial and secondarily generalized tonic-clonic seizures. N Engl J Med. 1985 Jul 18;313(3):145-51. doi: 10.1056/NEJM198507183130303. PMID 3925335
- [Background] Mattson RH, Cramer JA, Collins JF. A comparison of valproate with carbamazepine for the treatment of complex partial seizures and secondarily generalized tonic-clonic seizures in adults. The Department of Veterans Affairs Epilepsy Cooperative Study No. 264 Group. N Engl J Med. 1992 Sep 10;327(11):765-71. doi: 10.1056/NEJM199209103271104. PMID 1298221
- [Background] Mattson RH, Cramer JA, Collins JF. Prognosis for total control of complex partial and secondarily generalized tonic clonic seizures. Department of Veterans Affairs Epilepsy Cooperative Studies No. 118 and No. 264 Group. Neurology. 1996 Jul;47(1):68-76. doi: 10.1212/wnl.47.1.68. PMID 8710127
- [Background] Schmidt D. The clinical impact of new antiepileptic drugs after a decade of use in epilepsy. Epilepsy Res. 2002 Jun;50(1-2):21-32. doi: 10.1016/s0920-1211(02)00065-7. PMID 12151114
- [Background] Lhatoo SD, Wong IC, Polizzi G, Sander JW. Long-term retention rates of lamotrigine, gabapentin, and topiramate in chronic epilepsy. Epilepsia. 2000 Dec;41(12):1592-6. doi: 10.1111/j.1499-1654.2000.001592.x. PMID 11114218
- [Background] Morris GL 3rd, Mueller WM. Long-term treatment with vagus nerve stimulation in patients with refractory epilepsy. The Vagus Nerve Stimulation Study Group E01-E05. Neurology. 1999 Nov 10;53(8):1731-5. doi: 10.1212/wnl.53.8.1731. PMID 10563620
- [Background] Malow BA, Edwards J, Marzec M, Sagher O, Ross D, Fromes G. Vagus nerve stimulation reduces daytime sleepiness in epilepsy patients. Neurology. 2001 Sep 11;57(5):879-84. doi: 10.1212/wnl.57.5.879. PMID 11552020
- [Background] Harden CL, Pulver MC, Ravdin LD, Nikolov B, Halper JP, Labar DR. A Pilot Study of Mood in Epilepsy Patients Treated with Vagus Nerve Stimulation. Epilepsy Behav. 2000 Apr;1(2):93-99. doi: 10.1006/ebeh.2000.0046. PMID 12609137
- [Background] Elger G, Hoppe C, Falkai P, Rush AJ, Elger CE. Vagus nerve stimulation is associated with mood improvements in epilepsy patients. Epilepsy Res. 2000 Dec;42(2-3):203-10. doi: 10.1016/s0920-1211(00)00181-9. PMID 11074193
- [Background] Clark KB, Naritoku DK, Smith DC, Browning RA, Jensen RA. Enhanced recognition memory following vagus nerve stimulation in human subjects. Nat Neurosci. 1999 Jan;2(1):94-8. doi: 10.1038/4600. PMID 10195186
- [Background] McLachlan RS, Sadler M, Pillay N, Guberman A, Jones M, Wiebe S, Schneiderman J. Quality of life after vagus nerve stimulation for intractable epilepsy: is seizure control the only contributing factor? Eur Neurol. 2003;50(1):16-9. doi: 10.1159/000070853. PMID 12824707
- [Background] Cramer JA, Ben Menachem E, French J. Review of treatment options for refractory epilepsy: new medications and vagal nerve stimulation. Epilepsy Res. 2001 Nov;47(1-2):17-25. doi: 10.1016/s0920-1211(01)00286-8. PMID 11673017
- [Background] Gilliam FG, Fessler AJ, Baker G, Vahle V, Carter J, Attarian H. Systematic screening allows reduction of adverse antiepileptic drug effects: a randomized trial. Neurology. 2004 Jan 13;62(1):23-7. doi: 10.1212/wnl.62.1.23. PMID 14718691
- [Result] Ryvlin P, Gilliam FG, Nguyen DK, Colicchio G, Iudice A, Tinuper P, Zamponi N, Aguglia U, Wagner L, Minotti L, Stefan H, Boon P, Sadler M, Benna P, Raman P, Perucca E. The long-term effect of vagus nerve stimulation on quality of life in patients with pharmacoresistant focal epilepsy: the PuLsE (Open Prospective Randomized Long-term Effectiveness) trial. Epilepsia. 2014 Jun;55(6):893-900. doi: 10.1111/epi.12611. Epub 2014 Apr 22. PMID 24754318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between February 2006 and July 2008 and was prematurely terminated by Cyberonics, Inc. due to a low enrollment rate and not as a result of a safety or efficacy signal. There were 9 screen failures out of 131 screened patients, leaving 122 patients who started the study and are described in the Participant Flow.
Pre-assignment Details: Patients were randomized in a 1:1 ratio to the Best Medical Practice With Adjunctive VNS Therapy study group or to the Best Medical Practice Without VNS Therapy study group. VNS Therapy is delivered by an implantable device similar to a pacemaker that sends mild stimulation to the left vagus nerve to help improve seizure control.
Groups:
- Best Medical Practice: Best Medical Practice Without VNS Therapy
Period: Overall Study
Arm/Group | VNS Therapy | Best Medical Practice
Started | 59 | 63
Safety Set | 54 (Data of 5 randomized patients removed due to lack of ICF approval by site's local ethics committee.) | 58 (Data of 5 randomized patients removed due to lack of ICF approval by site's local ethics committee.)
Efficacy Set | 48 (6 pts. data excluded: exited prior to collection of baseline data & one postbaseline followup QOLIE) | 48 (10 pts. data excluded: exited prior to collection of baseline data & one postbaseline followup QOLIE)
Baseline and Month 3 | 47 (Completed Baseline and Month 3) | 47 (Completed Baseline and Month 3)
Baseline and Month 6 | 38 (Completed Baseline and Month 6) | 45 (Completed Baseline and Month 6)
Baseline and Month 9 | 33 (Completed Baseline and Month 9) | 35 (Completed Baseline and Month 9)
Baseline and Month 12 | 31 (Completed Baseline and Month 12) | 29 (Completed Baseline and Month 12)
Completed | 2 (Completed 2-year follow-up) | 5 (Completed 2-year follow-up)
Not Completed | 57 | 58
Not completed — Local IRB Consent Violation | 5 | 5
Not completed — Early Study Termination | 46 | 47
Not completed — Noncompliance | 2 | 2
Not completed — Reason Not Specified | 3 | 1
Not completed — Consent Withdraw | 1 | 2
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who completed the baseline assessment and at least one postbaseline follow-up QOLIE-89 assessment, and met local IRB consent requirements
Groups:
- Total: Total of all reporting groups
Arm/Group | VNS Therapy | Best Medical Practice | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Randomization
  Years | 38 (13) | 41 (11) | 40 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 24 | 27 | 51
Age of Epilepsy Onset [Mean (Standard Deviation); unit: years] | 13 (14) | 16 (14) | 15 (14)
Etiology of Epilepsy [Number; unit: participants]
  Structural/Metabolic | 26 | 26 | 52
  Unknown | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Quality of Life in Epilepsy-89 (QOLIE-89) Score in Patients With Baseline & at Least One Post-baseline QOLIE Assessment
Description: QOLIE-89 contains 17 multi-item measures of overall quality of life, emotional well-being, role limitations due to emotional problems, social support, social isolation, energy/fatigue, worry about seizure, medication effects, health discouragement, work/driving/social function, attention/concentration, language, memory, physical function, pain, role limitations due to physical problems, and health perceptions. Range of values 0-100. Higher scores reflect better quality of life; lower ones, worse quality of life.
Time Frame: Mean change from baseline QOLIE-89 Overall Score at 12 months
Population: Due to early study termination & only a few patients (n=7) achieving 2 year follow-up, study data for the 24 month time point is not available. However, at the 12 month time point there was an adequate amount of patient study data for analysis. This outcome measure evaluates the data for sixty (60) patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 31 | 29
units on a scale | 5.5 (7.2) | 1.2 (6.9)
Statistical Analysis 1: Comparison: VNS Therapy vs Best Medical Practice; Test type: Superiority or Other; p = .01, F Test

2. Secondary Outcome: Response Rate
Description: Response Rate is defined as the percent of participants who are responders. A Responder is defined as participants with a reduction of at least 50% or 75% in seizure frequency from baseline to the seizure count evaluation period.
Time Frame: Number of Responders at 12 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 31 | 29
participants | 10 | 7

3. Secondary Outcome: Percent of Patients That Are Seizure Free
Description: Percent of patients that are seizure free as defined by no seizures during the preceding follow-up period.
Time Frame: 3, 6, 9, 12, 15, 18, 21, 24 months
Population: This study was conducted between February 2006 and July 2008 and was prematurely terminated by Cyberonics, Inc. due to a low enrollment rate and not as a result of a safety or efficacy signal. Because of early termination and limited data this outcome measure was not tabulated.
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Percent Change in Seizure Frequency
Description: Percent change in total seizuires per week from baseline at 12 months
Time Frame: Mean percent change from baseline in seizure frequency at 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 31 | 29
Percent Change | -19.1 (43.92) | -1.0 (56.66)
Statistical Analysis 1: Comparison: VNS Therapy vs Best Medical Practice; Test type: Superiority or Other; p = 0.17, F-Test

5. Secondary Outcome: Seizure Free Days
Description: Seizure free days is defined as the time from last seizure to study exit date.
Time Frame: From the patient's last seizure to the study exit date
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Seizure Free Days Over the Last 6 Months
Time Frame: Over the last 6 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Center for Epidemiologic Studies Depression Scale (CES-D) Score
Description: The Center for Epidemiologic Studies Depression Scale (CES-D) includes 20 items comprising six scales reflecting major dimensions of depression: depressed mood, feelings of guilt and worthlessness, feelings of helplessness and hopelessness, psychomotor retardation, loss of appetite, and sleep disturbance. Possible range of scores is 0 to 60, higher scores indicate more depressive symptoms.
Time Frame: Mean change from baseline CES-D Score at 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 31 | 29
Units on a Scale | -2.2 (7.0) | 0.5 (8.1)
Statistical Analysis 1: Comparison: VNS Therapy vs Best Medical Practice; Test type: Superiority or Other; p = 0.17, F-Test

8. Secondary Outcome: Change From Baseline in Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) Score
Description: The Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) is a 6-item questionnaire validated to screen for depression in people with epilepsy. Scores range from 6 to 24, with higher scores indicating more depressive symptoms.
Time Frame: Mean change from baseline NDDI-E Score at 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 31 | 29
Units on a Scale | -1.0 (2.2) | -0.2 (3.4)
Statistical Analysis 1: Comparison: VNS Therapy vs Best Medical Practice; Test type: Superiority or Other; p = 0.28, F-Test

9. Secondary Outcome: Mean Change From Beginning of Intervention Clinical Global Impression-Improvement Scale (CGI-I) Score at 12 Months
Description: The Clinical Global Impression scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention Scores range from 1-7: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Mean change from baseline CGI-I Score at 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 31 | 29
Units on a Scale | -0.8 (0.8) | -0.3 (1.1)
Statistical Analysis 1: Comparison: VNS Therapy vs Best Medical Practice; Test type: Superiority or Other; p = 0.03, F-Test

10. Secondary Outcome: Change From Baseline in Adverse Event Profile (AEP) Score
Description: Adverse Events Profile (AEP) is a 19-item scale used as a systematic measure of adverse effects from antiepileptic drugs (AEDs). Scores range from 19-76; higher scores indicate high prevelance and severity of adverse events.
Time Frame: Mean change from baseline AEP Score at 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 31 | 29
Units on a scale | -6.0 (11.4) | -3.2 (6.9)
Statistical Analysis 1: Comparison: VNS Therapy vs Best Medical Practice; Test type: Superiority or Other; p = 0.26, F-Test

11. Secondary Outcome: Changes in Anti-epileptic Drugs (AEDs)
Description: Change from baseline in number of AED medications by visit
Time Frame: Change from baseline in number of AEDs at 12 months
Population: Due to early study termination & only a few patients (n=7) achieving 2 year follow-up, study data for the 24 month time point is not available. However, at the 12 month time point there was an adequate amount of patient study data for analysis. This outcome measure evaluates the data for fifty-nine (59) patients.
Measure: Median (Full Range); unit: Number of AEDs Taken
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 31 | 28
Number of AEDs Taken | 0 [-1 to 1] | 0 [-1 to 2]

12. Secondary Outcome: Retention Rate
Description: Percent of participants who were compliant with the protocol.
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Treatment Emergent Adverse Events, Device Complications, and Premature Study Withdrawal
Description: Number of participants with treatment emergent adverse events, device complications, and premature Study withdrawal.
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Quality of Life in Epilepsy - 89 Items(QOLIE-89)in Patients With Less Than a 50% Reduction in Seizures
Description: as for outcome 1
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Centre for Epidemiologic Studies Depression Scale (CES-D) in Patients With Less Then a 50% Reduction
Description: as for outcome 7
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) in Patients With Less Then a 50% Reduction in Seizures
Description: as for outcome 8
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Adverse Event Profile (AEP) in Patients With Less Then a 50% Reduction in Seizures
Description: as for outcome 10
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change in the Number of Anti-epileptic Drugs Prescribed
Description: Changes in Anti-Epileptic Drugs (AEDs) in patients with less then a 50% reduction in seizures
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Percent of Participants Who Were Compliant With the Protocol
Description: Retention rate in patients with less then a 50% reduction in seizures
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in QOLIE-89 Measures: Subgroup Analysis of Population With Baseline Adverse Event Profile Score >= 40
Description: QOLIE-89 contains 17 multi-item measures of overall quality of life. Range of values 0-100. Higher scores reflect better quality of life; lower ones, worse quality of life. Adverse Events Profile (AEP) is a 19-item scale used as a systematic measure of adverse effects from antiepileptic drugs (AEDs). Scores range from 19-76; higher scores indicate high prevelance and severity of adverse events.
Time Frame: Change from baseline up to 12 months
Population: This outcome measure includes patients from both arms, VNS + BMP (N=30) and BMP alone (N=31), with an overall QOLIE-89 at baseline and any other post baseline visit up to 12 months. Subgroup Analysis of population with Baseline Adverse Event Profile Score >= 40
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Groups:
- Baseline Adverse Event Profile Score >= 40: Population with Baseline Adverse Event Profile Score >= 40
Arm/Group | Baseline Adverse Event Profile Score >= 40
Number analyzed (Participants) | 61
Units on a Scale
  VNS Therapy | 3.3 (1.14)
  Best Medical Practice | 0.7 (1.08)

21. Secondary Outcome: Change From Baseline in QOLIE-89 Measures: Subgroup Analysis of Population With Baseline Adverse Event Profile Score < 40
Description: as for outcome 20
Time Frame: Change from baseline up to 12 months
Population: This outcome measure includes patients from both arms VNS + BMP (N=17) and BMP alone (N=17), with an overall QOLIE-89 at baseline and any other baseline visit up to 12 months. Subgroup Analysis of Population With Baseline Adverse Event Profile Score < 40
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Baseline Adverse Event Profile Score < 40: Population with Baseline Adverse Event Profile Score < 40
Arm/Group | Baseline Adverse Event Profile Score < 40
Number analyzed (Participants) | 34
units on a scale
  VNS Therapy | 3.3 (1.50)
  Best Medical Practice | 0.5 (1.52)

22. Secondary Outcome: Clinical Global Impressions Scale (CGI) in Patients With Less Then a 50% Reduction in Seizures
Description: The Clinical Global Impression scale (CGI-I)is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention Scores range from 1-7: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: At 12 and 24 months
Population: as for outcome 3
Arm/Group | VNS Therapy | Best Medical Practice
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: A total of 122 patients were randomized to receive VNS + BMP or BMP alone. Data from one study site (including 10 randomized patients) was removed from the analysis datasets due to lack of ICF approval by site's local ethics committee. The remaining 112, VNS + BMP (n=54) & BMP alone (n=58), randomized patients were included in the safety analyses.
Arm/Group | VNS Therapy | Best Medical Practice
Serious Adverse Events (participants affected / at risk) | 5/54 | 3/58
Other Adverse Events (participants affected / at risk) | 21/54 | 10/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS Therapy (N=54) | Best Medical Practice (N=58)
Depression (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 0 (0)
Suicide Attempt (General disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Prostate Cancer (Surgical and medical procedures) | 1 (2) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal Stone Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal Cord Paralysis (Nervous system disorders) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS Therapy (N=54) | Best Medical Practice (N=58)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 3 (3) | 0 (0)
Headache (General disorders) | 3 (3) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Eyelid Disorder (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Complication of Device Insertion (General disorders) | 1 (1) | 0 (0)
Facial Pain (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Localized Infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoesthesia (Nervous system disorders) | 3 (4) | 0 (0)
Mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Behavior (Psychiatric disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scar Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vocal Cord Paralysis (Nervous system disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated as a result of a decision by Cyberonics, Inc. The decision to terminate the study was primarily due to insufficient enrollment. The decision was not the result of a safety or efficacy signal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and Site agree not to publish or otherwise publicaly disclose clinical data generated in connection with the Study, unless approved in advance in writing by Cyberonics. Investigators and Site agree to provide Cyberonics with a copy of any proposed publication, abstract, or presentation relating to the research conducted under this Agreement at least 30 days prior to submission for publication or presentation.